CLINICAL TRIAL: NCT01536327
Title: Biomarker for Metachromatic Leukodystrophy Disease AN INTERNATIONAL, MULTICENTER, EPIDEMIOLOGICAL PROTOCOL
Brief Title: Biomarker for Metachromatic Leukodystrophy (BioMeta) Disease
Acronym: BioMeta
Status: Withdrawn | Type: Observational
Why Stopped: Transitioned to BioMetabol
Sponsor: CENTOGENE GmbH Rostock (Industry)
Responsible Party: Sponsor
Other Study IDs: BMLD 06-2018
Record Dates: First submitted 2012-02-21; First posted 2012-02-22 (Estimated); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Peripheral Neuropathy; Muscle Weakness
Keywords: leukodystrophies; Metachromatic Leukodystrophy Disease
MeSH Terms: conditions — Peripheral Nervous System Diseases; Muscle Weakness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — For the development of the new biomarkers using the technique of mass-spectometry, 10 ml EDTA blood sample and/or a dry blood spot filter card-blood sample will be taken from the patient. To prove the correct Metachromatic Leukodystrophy diagnosis in those patients where up to the enrolment in the study no genetic testing has been done, sequencing of Metachromatic Leukodystrophy will be done as routine diagnostic.
  The analyses will be done at the:
  Centogene AG Am Strande 7 18055 Rostock Germany
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Patients with Metachromatic Leukodystrophy disease or profound suspicion for Metachromatic Leukodystrophy disease

SUMMARY:
Development of a new MS-based biomarker for the early and sensitive diagnosis of Metachromatic Leu-kodystrophy disease from blood (plasma)

DETAILED DESCRIPTION:
Metachromatic Leukodystrophy Disease (MLD) is one of a group of genetic disorders called the leukodystrophies. These diseases impair the growth or development of the myelin sheath, the fatty covering that acts as an insulator around nerve fibers. Myelin, which lends its colour to the white matter of the brain, is a complex substance made up of varying lipids (75%) and proteins (25%). The leukodystrophies are caused by genetic defects in myelin production or metabolization of the compounds of the myelin sheath. Each of the leukodystrophies is the result of a defect in the gene that controls one (and only one) of the enzymes responsible for creating or degrading a part of the myelin. MLD is caused by a deficiency of the enzyme arylsulfatase A. MLD is one of several lipid storage diseases, which results in the toxic build-up of fatty materials (lipids) in cells in the nervous system, liver, and kidneys. There are three forms of MLD: late infantile, juvenile, and adult. Onset of the late infantile form (the most common MLD) is typically between 12 and 20 months following birth. Affected children have difficulty walking after the first year of life. Symptoms include muscle wasting and weakness, muscle rigidity, developmental delays, progressive loss of vision leading to blindness, convulsions, impaired swallowing, paralysis, and dementia. Children may become comatose. Most children with this form of MLD die by age 5. The juvenile form of MLD (between 3-10 years of age) usually begins with impaired school performance, mental deterioration, and dementia and then develop symptoms similar to the infantile form but with slower progression. The adult form commonly begins after age 16 as a psychiatric dis-order or progressive dementia. Symptoms include impaired concentration, ataxia, seizures, dementia, and tremor. Due to consanguinity autosomalrecessive disorders such as MLD have higher prevalence in Arabian countries.

New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood (plasma) of affected patients that allow to diagnose in the future the disease earlier, with a higher sensitivity and specificity. In a pilotstudy glycosylsphingosin-sulfatid has been determined as a sensitive and specific biomarker. This is a metabolic product likely to be involved in the pathophysiology of the disease. Therefore it is the goal of the study to validate this new biochemical marker from the blood (plasma) of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment. Examining blood samples will allow to determine whether measurement of the identified marker lyso-Gb1-Sulfatid is feasible in blood samples and will further promote early detection of MLD.

Though MLD is a pan-ethnic disorder, the prevalence of this autosomal-recessive disorder is elevated in countries with a higher frequency of consanguinity. Therefore, we estimate that every 400th newborn in Arabian countries may be eligible for inclusion due to high-grade suspicion of MLD, while approximately every 2000th newborn in a non-Arabian country may be eligible.

ELIGIBILITY:
INCLUSION CRITERIA:

* Informed consent will be obtained from the patient or the parents before any study related procedures
* Patients from one day
* The patient has a diagnosis of Metachromatic Leukodystrophy disease or profound suspicion for Metachromatic Leukodystro-phy disease
* High-grade suspicion present, if one or more criteria are valid:

Positive family anamnesis for MLD

Neurologic symptoms of unknown origin: peripheral neuropathy, clumsiness, choreatiform movements, spastic quadriplegia, loss of ambulation, bulbar dysfunction/paresis, dysphagia, seizure disorders

Psychiatric symptoms of unknown origin: mental regression, emotional la-bility, disorganized thinking or hallucinations/delusions

Muscle symptoms of unknown origin: muscle weakness

EXCLUSION CRITERIA:

* No Informed consent from the patient or the parents before any study related procedures
* No diagnosis of MLD or no valid criteria for high-grade suspicion of MLD

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Metachromatic Leukodystrophy disease or profound suspicion for Metachromatic Leukodystrophy disease
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-08-20 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-02-28 (Actual)

PRIMARY OUTCOMES:
Development of a new MS-based biomarker for the early and sensitive diagnosis of metachromatic leukodystrophy disease from the blood | 24 month
  New methods, like mass-spectrometry give a good chance to characterize specific metabolic alterations in the blood of affected patients that allow diagnosing in the future the disease earlier, with a higher sensitivity and specificity.

SECONDARY OUTCOMES:
Testing for clinical robustness, specificity and long-term stability of the biomarker | 36 months
  the goal of the study to identify and validate a new biochemical marker from the blood of the affected patients helping to benefit other patients by an early diagnose and thereby with an earlier treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Bauer, Prof., Study Chair — Centogene GmbH
Locations (5):
- Children's Hospital, Faculty of Medicine, Ain Shams University, Cairo, Egypt
- Centogene AG, Rostock, Germany
- India (2):
  - Amrita Institute of Medical Sciences & Research Centre, Kochi, Kerala
  - Navi Mumbai Institute of Research In Mental And Neurological Handicap (NIRMAN), Mumbai
- Lady Ridgeway Hospital for Children, Colombo, Sri Lanka

IPD SHARING:
Plan to Share IPD: No